CLINICAL TRIAL: NCT06098924
Title: The Impacts of Spiritual Health on Depression and Happiness Among Hemodialysis Patients: the Moderator Effects of Life-meaning and Post-trauma Growth
Brief Title: HD Patients' Depression and Happiness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ya-Chu Hsiao, professor, Chang Gung University of Science and Technology
Other Study IDs: NSCT-112-2014-H-255-009
Record Dates: First submitted 2023-10-15; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Hemodialysis
Keywords: spirituality; depression; happiness; post-trauma growth; life meaning
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to verify the mediating effect of life of meaning and post-traumatic growth in spirituality and psychological well-being (happiness, depression).

DETAILED DESCRIPTION:
The research design is cross-sectional correlational study. Convenient sampling will be used to conduct to data collection. There are 300 patients with hemodialysis from a hemodialysis institution in the north Taiwan, and data collecting with self-administrated questionnaires. The instruments include demographic and disease-related information, Spiritual Health Scale short form, Chinese Happiness Inventory, Beck Depression Inventory-II, Life Attitude Profile, Posttraumatic Growth Inventory. The SPSS 22.0 statistical software will be used to analyze the data. Descriptive statistics, such as frequency, percentage, mean, and standard deviation (SD) will be used for participant characteristics and outcome measures. T-test, chi-square, ANOVA, post-hoc, ANCOVA, and Person's correlation will be conducted to test the relationships between the research variables.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are over 20 years old
* voluntarily participate in the study and sign the respondent consent form
* have received routine hemodialysis treatment for more than three months
* have clear consciousness and can communicate in Mandarin and Taiwanese.

Exclusion Criteria:

* Patients whose medical records record a diagnosis of schizophrenia
* patients are taking antidepressant drugs

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with regularly hemodylysis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The status of spirituality among HD patients | 1 day
  Self-administrated questionnaire of Spiritual Health Scale short form was used to collect data. The score range is 24 to 120, and the higher score means higher spirituality.
The status of life-meaning among HD patients | 1 day
  Self-administrated questionnaire of Life Attitude Profile was used to collect data. The score range is 39 to 195, and the higher score means higher level of life-meaning.
The status of post-trauma growth among HD patients | 1 day
  Self-administrated questionnaire of Posttraumatic Growth Inventory was used to collect data. The score range is 0 to 105, and the higher score means higher level of post-trauma growth.
The status of depression among HD patients | 7 minutes
  Self-administrated questionnaire of Beck Depression Inventory-II was used to collect data. The score range is 0 to 63, and the higher score means higher level of depressive tendency.
The status of happiness among HD patients | 1 day
  Self-administrated questionnaire of Chinese Happiness Inventory was used to collect data. The score range is 0 to 30, and the higher score means higher level of happiness.
The mediating effect of life of meaning and post-traumatic growth | 1 day
  Using these scores form these scales (mention above) to verify the mediating effect of life of meaning and post-traumatic growth in spirituality and psychological well-being (including happiness, depression).

CONTACTS AND LOCATIONS:
Overall Officials: yachu hsiao, Principal Investigator — Chang Gung University of Science and Technology
Locations (1):
- Chang Gung University of Science and Technology, Taoyuan, N/A = Not Applicable, Taiwan

IPD SHARING:
Plan to Share IPD: No